CLINICAL TRIAL: NCT02108522
Title: Administration of Most Closely HLA-matched Multivirus-specific Cytotoxic T-Lymphocytes for the Treatment of EBV, CMV, Adenovirus, HHV6, and BK Virus Infections Post Allogeneic Stem Cell Transplant
Brief Title: Multivirus-specific T Cells for the Treatment of Virus Infections After Stem Cell Transplant
Acronym: CHARMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AlloVir (Industry)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-33903, CHARMS
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Infection
Keywords: CMV infection; EBV infection; HHV6 virus infection; BK virus infection; Adenovirus infection; JC virus infection; allogeneic stem cell transplant; Virus Specific T cells
MeSH Terms: conditions — Infections; Cytomegalovirus Infections; Epstein-Barr Virus Infections; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multivirus Specific T cells (Experimental): Partially HLA-matched multivirus specific T cells (VSTs) will be thawed and given by intravenous injection. Patients will receive 2 x 10^7 VSTs/m2 as a single infusion. In the rare case where insufficient banked cell product is available, a lower number of cells may be infused after discussion with the principal investigator, patient and/or guardian and the treatment team.
  If after the first treatment there is persistent infection, there is an option to receive more treatments. These additional treatments might be with cells from the same donor or another donor whose cells are also thought to be a good match for the patient and effective against their virus. This second product will be administered at the same dose level 28 days after the initial infusion, and subsequent infusions should be at least 14 days apart.
  Interventions: Biological: Multivirus Specific T cells

INTERVENTIONS:
Biological: Multivirus Specific T cells

SUMMARY:
Patients enrolled on this study will have received a stem cell transplant. After a transplant, while the immune system grows back the patient is at risk for infection. Some viruses can stay in the body for life and if the immune system is weakened, like after a transplant, they can cause life threatening infections.

Patients enrolled on this study will have had an infection with one or more of the following viruses - Epstein Barr virus (EBV), cytomegalovirus (CMV), BK virus, JC virus, adenovirus or HHV6 (Human Herpes Virus 6).

Investigators want to see if they can use a kind of white blood cell called T cells to treat infections of these viruses after a transplant. Investigators have observed in other studies that treatment with specially trained T cells has been successful when the cells are made from the transplant donor. However as it takes 1-2 months to make the cells, that approach is not practical when a patient already has an infection.

Investigators have now generated multivirus-specific T cells (VSTs) from the blood of healthy donors and created a bank of these cells. Investigators have previously successfully used frozen multivirus-specific T cells from healthy donors to treat virus infections after bone marrow transplant and now have improved the production method to make it safer and target more viruses.

In this study, investigators want to find out if they can use these banked VSTs to fight infections caused by the viruses mentioned above.

DETAILED DESCRIPTION:
These VST lines have been made at Baylor College of Medicine from donors for other transplant patients or other normal donors some of whom were from the National Marrow Donor Program. All donors have been screened with the standard blood bank donor questionnaire, medical history and testing for infectious disease by a doctor who is experienced in screening transplant donors. Only donors who have cleared this process and were deemed to be eligible provided blood for VST generation.

The lines were made using a special process. To make the VSTs investigators mixed donor cells with small pieces of proteins, called peptides that come from adenovirus, CMV, EBV, BKV and HHV6. These peptides stimulate donor T cells that react against the viruses to grow and train the donor T cells to kill cells that are infected with CMV, EBV, adenovirus, BKV and HHV6.

Once the investigators made sufficient numbers of VSTs, they tested them to make sure they would target cells infected with these viruses but not normal cells. Then the cells were frozen.

For patients treated on this study, the VSTs will be thawed and injected into their intravenous line. The patient will remain in the clinic for at least one hour after the infusion. After the patient receives the cells, their transplant doctor will monitor the levels of the virus the patient is infected with in their blood. The investigators will also take blood to see how long the VSTs given to the patient last in their body.

The patient will continue to be followed by their doctors after the injection. The patient will either be seen in the clinic or will be contacted by a research nurse to follow up for this study every week for 6 weeks then at 3, 6 and 12 months. The patient may have other visits for their standard care.

The patient will also have regular blood tests done to follow their counts and the viral infection, but most of these will be done as part of their standard medical care. To learn more about the way the VSTs are working in the patient's body, up to an extra 30-40 ml (6-8 teaspoons) of blood will be taken before the infusion and then at 1, 2, 3, 4, 6 weeks and 3 months. Blood should come from the central intravenous line, and should not require extra needle sticks.

All participants on this study will be infused with the same number (dose) of cells. If after the first treatment the patient has a persistent infection, we would discuss this with him/her and allow an option to receive more treatments. These additional treatments might be with cells from the same donor or if we feel that there is another donor's whose cells might be better for the patient, we would use cells from a different donor. This second product will be administered at the same dose level 28 days after the initial infusion, and subsequent infusions should be at least 14 days apart. After each VST infusion, the patient will be monitored as described above.

ELIGIBILITY:
Inclusion Criteria:

For Initial VSTs and subsequent infusions: patients will be eligible following any type of allogeneic transplant if they have CMV, adenovirus, EBV, BK virus and/or HHV6 infection/disease persistent or recurrent despite 14 days of standard therapy OR after failure of treatment after 7 days of standard therapy OR if unable to tolerate standard therapy. Patients with persistent JC virus infection will be eligible as well.

1. Prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant using either bone marrow or peripheral blood stem cells or single or double cord blood.
2. Treatment of the following persistent or relapsed infections despite standard therapy;

   1. CMV: Treatment of persistent or relapsed CMV disease or infection after standard therapy. For CMV infection, standard therapy is defined as antiviral therapy with ganciclovir, foscarnet or cidofovir.

      * CMV disease: defined as the demonstration of CMV by biopsy specimen from visceral sites (by culture or histology) or the detection of CMV by culture or direct fluorescent antibody stain in bronchoalveolar lavage fluid in the presence of new or changing pulmonary infiltrates or changes consistent with CMV retinitis on ophthalmologic examination.
      * CMV infection: defined as the presence of CMV positivity as detected by PCR or pp65 antigenemia or culture from ONE site such as stool or blood or urine or nasopharynx.
      * Failure of antiviral therapy: defined as a rise or a fall of less than 50% in viral load in peripheral blood or any site of disease as measured by PCR or pp65 antigenemia after 7 days of antiviral therapy.
   2. Adenovirus: Treatment of persistent adenovirus infection or disease despite standard therapy. Standard therapy is defined as antiviral therapy with cidofovir or an alternative antiviral agent if patient will not tolerate cidofovir therapy because of poor renal function.

      * Adenovirus infection: defined as the presence of adenoviral positivity as detected by PCR or culture from ONE site such as stool or blood or urine or nasopharynx.
      * Adenovirus disease: defined as the presence of adenoviral positivity as detected by PCR, DFA or culture from two or more sites such as stool or blood or urine or nasopharynx.
      * Failure of therapy: defined as a rise or a fall of less than 50% in viral load in peripheral blood or any site of disease as measured by PCR or any other quantitative assay) after 7 days of antiviral therapy.
   3. EBV: For treatment of persistent EBV infection despite standard therapy. For EBV infection, standard therapy is defined as rituximab given at 375mg/m2 in patients for 1-4 doses with a CD20+ve tumor.

      * EBV infection: defined as Biopsy proven lymphoma with EBV genomes detected in tumor cells by immunocytochemistry or in situ PCR,Or clinical or imaging findings consistent with EBV lymphoma and/or elevated EBV viral load in peripheral blood.
      * Failure of therapy is defined as: Increase or less than 50% response at sites of disease for EBV lymphoma OR, Increase or a fall of less than 50% in EBV viral load in peripheral blood or any site of disease after 1st dose of rituximab.
   4. BK virus: Treatment of persistent BK virus infection or BK virus disease despite antiviral treatment with cidofovir or leflunomide. No clear standard treatment is defined. Cidofovir has been administered in low doses as well as high doses to HSCT patients with BK infections but no randomized trials are available proving its clinical efficacy. In small trials leflunomide had activity against BK virus, therefore we will consider this agent an acceptable alternative to cidofovir, given the absence of a clear first line option.

      * BK virus infection is defined as the presence of BK virus positivity as detected by PCR or culture in one site such as blood or urine.
      * BK virus disease is defined as the presence of BK virus detectable by culture or PCR in blood or urine or other body fluids and symptoms of disease including, but not limited to persistent microscopic or macroscopic hematuria or detectable BK virus in more than one site.
      * Failure of therapy is defined as a rise or a fall of less than 50% in viral load in peripheral blood or any site of disease as measured by PCR or any other quantitative assay) or worsening hematuria after 7 days of antiviral therapy.
   5. HHV6: Treatment of persistent HHV6 infection or disease despite antiviral treatment with ganciclovir, cidofovir and foscarnet. No clear standard treatment is defined. Ganciclovir, cidofovir and foscarnet all have variable in vitro activity against HHV-6, and may have a role in treating HHV-6-associated disease - therefore antiviral treatment with one or more of these agents will we acceptable initial therapy.

      * HHV6 virus infection is defined as the presence of elevated HHV-6 levels as detected by PCR or positive culture in one site such as CSF or blood.
      * HHV6 disease is defined as defined as the presence of HHV6 detectable by culture or PCR in one or more sites such as blood or CSF and symptoms of disease including symptoms of HHV6 encephalitis OR detectable HHV6 by PCR or culture in more than one site.
      * Failure of therapy is defined as a rise or a fall of less than 50% in viral load in peripheral blood or any site of disease (as measured by PCR or any other quantitative assay) after 7 days of antiviral therapy.
   6. JC virus: Treatment of progressive or persistent JC virus infection or disease without suitable alternative treatment option. Pepmixes specific for antigens on adenovirus, EBV, CMV, HHV6 and BK virus are used to generate our multivirus-specific VSTs. No pepmix specific for the rare JC virus is used for generation of these CTLs, however given the high homology (>90%) between JC and BK and the fact that BK virus-specific T cells targeting VP1 and Large T (as targeted in our multivirus VSTs) have been administered to treat JCV-PML, resulting in viral clearance from the cerebrospinal fluid it is likely that our VSTs are efficacious against JC virus. Given the current lack of treatment options for JC virus infection or reactivation after HSCT and the risk of progression to JML, which is almost uniformly fatal, and the apparent activity of BK virus-directed T cells against JC virus infected cells, we propose including patients with progressive or persistent JC virus on this study, unless a suitable alternative therapy is available.

      * JC virus infection is defined as the presence of elevated JC virus levels as detected by PCR or positive culture in one site such as CSF or blood.
      * JC virus disease is defined as defined as the presence of JC virus detectable by culture or PCR in one or more sites such as blood or CSF and symptoms of disease including symptoms of PML OR detectable JC virus by PCR or culture in more than one site.
3. Patients with multiple CMV, EBV, Adenovirus, HHV6 and BK virus infections are eligible given that each infection is persistent despite standard therapy as defined above. Patients with multiple infections with one or more reactivation and one or more controlled infection are eligible to enroll.
4. Clinical status at enrollment to allow tapering of steroids to equal or less than 0.5 mg/kg/day prednisone (or equivalent).
5. HgB>8.0
6. Pulse oximetry of > 90% on room air
7. Available multivirus-specific VSTs
8. Negative pregnancy test in female patients if applicable (childbearing potential who have received a reduced intensity conditioning regimen).
9. Written informed consent and/or signed assent line from patient, parent or guardian.

Exclusion Criteria:

1. Patients receiving ATG, Campath or other immunosuppressive T cell monoclonal antibodies within 28 days of screening for enrollment.
2. Patients with other uncontrolled infections. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment.

   Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
3. Patients who are less than 28 days removed from their allogeneic hematopoietic stem cell transplant or who have received donor lymphocyte infusions (DLI) within 28 days.
4. Patients with active acute GVHD grades II-IV.
5. Active and uncontrolled relapse of malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-06; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Omer, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Derived] Pfeiffer T, Tzannou I, Wu M, Ramos C, Sasa G, Martinez C, Lulla P, Krance RA, Scherer L, Ruderfer D, Naik S, Bocchini C, Fraser IP, Patel B, Ward D, Wang T, Heslop HE, Leen AM, Omer B. Posoleucel, an Allogeneic, Off-the-Shelf Multivirus-Specific T-Cell Therapy, for the Treatment of Refractory Viral Infections in the Post-HCT Setting. Clin Cancer Res. 2023 Jan 17;29(2):324-330. doi: 10.1158/1078-0432.CCR-22-2415. PMID 36628536

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigational product was administered to 58 unique patients. However, one patient was enrolled twice for two separate infections. An additional 24 patients were screened but did not receive investigational product.
Period: Screening Period
Arm/Group | Multivirus Specific T Cells
Started | 82
Completed | 58
Not Completed | 24
Period: Period 1: Initial Cohort
Arm/Group | Multivirus Specific T Cells
Started | 50
Completed | 28
Not Completed | 22
Period: Period 2: Expansion Cohort
Arm/Group | Multivirus Specific T Cells
Started | 8
Completed | 2
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: Investigational product was administered to 58 unique patients, however one patient was enrolled twice for two separate infections. An additional 24 patients were screened but did not receive investigational product.
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants] — Population: Age was not collected for patients who were screened for the study but did not receive investigational product.
  Participants
    <=18 years | 21
    Between 18 and 65 years | 33
    >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 33 [2 to 73]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographics for patients who were screened for the study but did not receive investigational product were not collected.
  Participants
    Female | 28
    Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 51
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Where a Suitable VST Line Could be Found
Description: Consented subjects will be screened for a suitable VST line to asses feasibility of finding a sufficiently matching VST line.
Time Frame: within 24 hours of receiving recipient HLA information
Population: Includes all patients screened for the study
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 82
Participants | 80

2. Primary Outcome: Number of Patients With Acute GvHD Grades III-IV
Description: Safety of VSTs based on patients with acute GvHD grades III-IV within 42 days of the last dose of VSTs. Acute GVHD grading was performed by the consensus conference criteria (1). Grade 0 represents no acute GvHD. Grade 4 represents the most severe acute GvHD.
Time Frame: 42 days
Population: Includes all patients who received at least one dose of investigational product
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 58
Participants | 1

3. Primary Outcome: Number of Patients With Grades 3-5 Non-hematologic Adverse Events Related to the T Cell Product
Description: Safety of VSTs based on patients with grades 3-5 non-hematologic adverse events that are at least possibly related to the T cell product within 28 days of the last VST dose by NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Grade 1 Mild; asymptomatic or mild symptoms. Grade 2 Moderate symptoms. Grade 3 Severe or medically significant but not immediately life-threatening. Grade 4 Life-threatening consequences. Grade 5 Death related to AE.
Time Frame: 28 days
Population: Includes all patients who received at least one dose of investigational product. There were no patients with grade 5, 1 patient with grade 4, and 5 patients with grade 3 treatment related adverse experiences.
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 58
Participants | 6

4. Secondary Outcome: Number of Participants With a Viral Response at 42 Days
Description: Viral response is defined as follows: Complete response: Return to normal range as defined by specific assay used and clinical signs and symptoms. Partial response: Decrease in viral load of at least 50% from baseline or 50% improvement of clinical signs and symptoms.
Time Frame: 42 days
Population: Includes all patients who received at least one dose of investigational product
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 58
Participants | 54

5. Secondary Outcome: Number of Patients With Reconstitution of Antiviral Immunity (as Measured in Peripheral Blood)
Description: Reconstitution of Antiviral Immunity as detected during the study as defined by virus-specific T cells > 10 SFC/5x10e5 PBMCs for one virus or additive within the first 6 weeks after the first infusion. As determined by interferon-gamma ELISpot assay of PBMCs after stimulation with virus-specific peptides. Assay reflects antiviral activity in peripheral blood, not necessarily in the site of viral infection. Patients could therefore have a negative result in the presence of antiviral immunity.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 55
Participants | 28

6. Secondary Outcome: Persistence of VSTs (in Peripheral Blood)
Description: Number of patients with circulating T cells of confirmed 3rd party origin as measured by epitope mapping and other techniques. Infused versus endogenous cells were discriminated on the basis of peptide-epitope specificity in patients with adequate PBMC numbers and available reagents.
Time Frame: Within 6 weeks
Population: Includes only patients who had at least 1 dose of investigational product, and had cells collected for analysis within 6 weeks of infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 16
Participants | 11

7. Secondary Outcome: Association Between High HLA Matching and Viral Outcomes
Description: Patients with 4-8 matching alleles (high HLA match) and complete or partial viral response (Viral response is defined as follows: Complete response: Return to normal range as defined by specific assay used and clinical signs and symptoms. Partial response: Decrease in viral load of at least 50% from baseline or 50% improvement of clinical signs and symptoms). See Outcome Measure 8 for low-matching outcomes.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 21
Participants | 18

8. Secondary Outcome: Association Between Low HLA Matching and Viral Outcomes
Description: Patients with 1-3 matching alleles (low HLA match) and complete or partial viral response (Viral response is defined as follows: Complete response: Return to normal range as defined by specific assay used and clinical signs and symptoms. Partial response: Decrease in viral load of at least 50% from baseline or 50% improvement of clinical signs and symptoms.) See Outcome Measure 7 for high-matching outcomes.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 16
Participants | 16

9. Secondary Outcome: Number of Patients With a Clinical Response 3 Months After the First Dose of VSTs
Description: as for outcome 4
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 58
Participants | 54

10. Secondary Outcome: Number of Patients With Non-target Viral Reactivations Within 12 Months
Description: All CMV, EBV, adenovirus, BK virus, JC virus and HHV6 infections/reactivations, other than the primary infection, occurring within 12 months of VST infusion. These viral infections could have occurred after clearance of the infused VST.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 58
Participants | 19

11. Secondary Outcome: Number of Patients With Secondary Graft Failure at 30 Days
Description: Secondary graft failure is defined as initial neutrophil engraftment followed by subsequent decline in the ANC to less than 500/mm^3 for three consecutive measurements on different days, unresponsive to growth factor therapy that persists for at least 14 days in the absence of a known cause such as relapse. Population includes patients with serious adverse experiences potentially related to VSTs who did not have an alternative explanation for graft failure, such as disseminated tuberculosis, or toxicity of other therapies eg. ganciclovir.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 58
Participants | 0

12. Secondary Outcome: Number of Patients With Chronic GVHD
Description: Number of patients with new or worsened chronic GVHD by standard criteria. By standard criteria, overall severity of chronic GvHD could be scored as none, mild, moderate, or severe.
Time Frame: 12 months
Population: Includes all patients that were assessed for chronic GVHD. Eight patients had chronic GVHD. All 8 patients evaluated with chronic GVHD had either preexisting or a history of acute or chronic GVHD.
Measure: Count of Participants; unit: Participants
Arm/Group | Multivirus Specific T Cells
Number analyzed (Participants) | 36
Participants | 8

ADVERSE EVENTS:
Time Frame: From first injection of study drug up to 28 days after last injection of study drug
Description: Non-hematologic adverse events, grades 3-5 (according to common terminology criteria for adverse events)
Arm/Group | Multivirus Specific T Cells
All-Cause Mortality (participants affected / at risk) | 6/58
Serious Adverse Events (participants affected / at risk) | 17/58
Other Adverse Events (participants affected / at risk) | 15/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multivirus Specific T Cells (N=58)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Aspartate Aminotransferase Increased (Hepatobiliary disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 2 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Platelet Count Decreased (Blood and lymphatic system disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Multi-organ failure (General disorders) | 3 (3)
Nausea (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Renal Failure (Hepatobiliary disorders) | 1 (1)
Coronavirus Infection (Infections and infestations) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine Increased (Investigations) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multivirus Specific T Cells (N=58)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Abdominal Pain (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 5 (5)
Pyrexia (General disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Limited information is available regarding patients who were screened for the study but were not administered investigational product. Data are preliminary and unaudited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT02108522/Prot_SAP_000.pdf